CLINICAL TRIAL: NCT03777722
Title: Light, Metabolic Syndrome and Alzheimer's Disease: A Non-Pharmocological Approach
Brief Title: Light and the Effect on Metabolic Syndrome and Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Rutgers University (Other)
Responsible Party: Principal Investigator, Mariana Figueiro, Professor, Population Health Science and Policy, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 17-2685
Record Dates: First submitted 2018-12-12; First posted 2018-12-17 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Alzheimer Disease; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Crossover placebo controlled design
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aim 1: Active Intervention then Placebo (Experimental): Tailored Lighting intervention (TLI). The active TLI will provide high circadian stimulation during the day produced by light sources that provide moderate light levels of spectra that are tuned to the sensitivity of the circadian system. The active lighting intervention will be in place for 8 weeks. Following an 8 week washout period, the participants will see the placebo control intervention for 8 weeks.
  Interventions: Device: Tailored Lighting Intervention
- Aim 1: Placebo Intervention then Active (Experimental): The placebo lighting intervention is designed to have no effect on the circadian system. The control intervention will be in place for 8 weeks. Following an 8 week washout period, the participants will see the active tailored lighting intervention for 8 weeks.
  Interventions: Device: Tailored Lighting Intervention

INTERVENTIONS:
Device: Tailored Lighting Intervention — Lighting Intervention - active or placebo

SUMMARY:
This study's main hypothesis is that a delivering a tailored lighting intervention (TLI) will provide a successful means for promoting circadian entrainment and treating metabolic disease and inflammation in patients with mild cognitive impairment (MCI) and Alzheimer's disease (AD) and Alzheimer's disease and related dementias (ADRD). As such, the proposed studies have the potential to provide important insights into the link between AD/ADRD and type 2 diabetes (T2DM) by identifying the disruption of circadian rhythms as a key component in the metabolic impairment. Preliminary data from ongoing studies demonstrates a beneficial effect of light treatment on sleep and depression. If positive results are observed, the potential also exists to transform the manner in which homes, assisted living facilities, and nursing homes are lighted by delivering a simple, practical, non-pharmacological intervention to promote entrainment, improve sleep, and reduce metabolic disease in AD and mild AD MCI patients. This randomized, placebo-controlled, crossover study involving 60 AD/ADRD patients who live in controlled environments (i.e., assisted living facilities and nursing homes), will investigate whether 8 weeks of exposure to a TLI designed to increase circadian entrainment improves sleep, mood, inflammatory markers, and metabolic control, compared to a control, circadian-inactive light.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) and type 2 diabetes (T2DM) pose linked, major threats to aging societies worldwide, but the relationship between these two diseases remains poorly understood. Hence, insulin resistance may account for the close epidemiological association between AD and T2DM. A major gap in the understanding of this association, however, is how brain insulin resistance develops in the context of AD. Studies show that circadian disruption impairs metabolic control and increases the risk for diabetes and obesity. Vice versa, disrupted sleep and depression are closely linked to impaired metabolic control and increased diabetes risk in the general population. Notably, AD is associated with circadian disruption, which may be amplified by exposure to irregular light-dark patterns or constant dim light. To what extent circadian disruption contributes to increased diabetes risk in AD remains unclear. Here, the investigator aims to test whether a novel tailored lighting intervention (TLI) designed to promote circadian entrainment in AD patients can improve metabolic control. Preliminary data from ongoing studies demonstrates a beneficial effect of light treatment on sleep and depression. Given the close association of sleep on metabolic control, these data support the hypothesis that light therapy that promotes entrainment can restore metabolic control in AD patients. Specifically, the investigator will test the efficacy of a practical, scientifically sophisticated 24-hour lighting system for increasing circadian entrainment in older adults with AD and related dementias (ADRD). The major goal is to demonstrate that a practical, effective, tailored, nonpharmacological intervention that promotes circadian entrainment can be used to improve sleep, reduce inflammation, and ameliorate glucose intolerance and insulin resistance in AD/ADRD patients.

Aim 1: Test if a TLI that promotes entrainment can improve sleep, depression, inflammation, and glucose tolerance in patients with moderate to late stages ADRD. In a randomized, placebo-controlled, crossover study involving 60 ADRD patients who live in controlled environments, the investigators will investigate whether an 8-week exposure to a TLI designed to increase circadian entrainment (urinary melatonin and activity-rest patterns) will improve inflammation and glucose tolerance (oral glucose tolerance test), and reduce sleep disturbances (actigraphy, Pittsburgh Sleep Quality Index, PSQI) and depressive symptoms (Cornell Scale for Depression in Dementia, CSDD) compared to a control, circadian-inactive light.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild to moderate Alzheimer's disease or related dementia,
* sleep disturbance as determined by a score ≥ 5 on the PSQI

Exclusion Criteria:

* insulin-dependent diabetes,
* urinary incontinence
* obstructing cataracts
* macular degeneration
* blindness
* severe sleep apnea or
* restless leg syndrome (RLS)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Glucose tolerance | once during weeks 1 (baseline), 5, 9, 18 (second baseline), 22, and 26
  change in glucose tolerance from baseline will be assessed using an oral glucose tolerance test

SECONDARY OUTCOMES:
Sleep Efficiency using actigraphy | 7 days during weeks 1 (baseline), 5, 9, 18 (second baseline), 22, and 26
  Actigraphs will be worn for 7 days during assessment weeks. Actigraphy will be used to calculate changes in sleep efficiency. A higher sleep efficiency indicates better sleep.
Light exposure using the Daysimeter | 7 days during weeks 1 (baseline), 5, 9, 18 (second baseline), 22, and 26
  Daysimeters will be worn for 7 days during assessment periods to measure the amount of circadian effective light delivered by the lighting intervention.
Change in sleep disturbance | once during weeks 1 (baseline), 5, 9, 18 (second baseline), 22, and 26
  Change in sleep disturbance will be assessed using the Pittsburgh Sleep Quality Index. The sum of the 7 component scores yields a single global score. A person with a global score above 5 is considered to have sleep disturbances. A higher score indicates worsening sleep disturbance.
Change in depression | once during weeks 1 (baseline), 5, 9, 18 (second baseline), 22, and 26
  A change in depression will be assessed using the Cornell Scale for Depression in Dementia. A score of twelve or more points indicates depression. A higher score indicates worsening depression.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Figueiro, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Rutgers University, New Brunswick, New Jersey
  - Icahn School of Medicine at Mount Sinai, Albany, New York
  - Icahn School of Medicine, New York, New York